CLINICAL TRIAL: NCT03666936
Title: A Social-Healthcare Pathway to Facilitate Return to Work of Cancer Survivors in Italy: Implementation Process of the UNAMANO Project
Brief Title: Facilitate the Return to Work of Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCCA_Welcom_2017
Record Dates: First submitted 2018-08-20; First posted 2018-09-12 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2021-07

CONDITIONS: Neoplasms; Return to Work
Keywords: Cancer survivors; Return to work; Italy; Occupational Therapy; Comprehensive Health Care; Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Social-health care intervention
  Interventions: Other: Social-health care intervention

INTERVENTIONS:
Other: Social-health care intervention — Cancer survivors enrolled in the study could receive support from the Occupational Therapist and/or from the social care professionist to overcome the difficulties encounter at work or to facilitate work reintegration.

SUMMARY:
Cancer patients could experience physical limitations, cognitive symptoms, fatigue and pain, that could be perceived at diagnosis but may also occur during treatment, limiting the person from carrying out their activities of daily living, including work tasks. Return to work is a major goal, as it facilitates the patient's ability to deal with the disease and improve general health.

At present, there is no path aimed at supporting cancer patients in the return to work process. Because of this, the investigators want to assess the feasibility of a multidisciplinary social-health care pathway aimed at manage the difficulties that cancer patients might perceive in the return to work process.

DETAILED DESCRIPTION:
To receive the support from the social-health care pathway, cancer survivors should go to an information desk service (called Informa Salute) located in the hospital. Here, sociodemographic and work-related data will be collected with the aim to organize the tailored social-health support to facilitate the return to work.

The social-health care pathway created includes: the local Health Authority of Reggio Emilia and the local Order of Physicians, voluntary non-profit associations, vocational and educational training bodies, social cooperatives, one labor union and one chartered accountant enterprise.

ELIGIBILITY:
Inclusion Criteria:

* adults with cancer diagnosis and employed at the time of diagnosis

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
number, type and duration of intervention provided (information, occupational therapy, social support) and, for those who have been offered the involvement of the employer, the number of those who have accepted this intervention (Feasibility indicator_1) | through study completion, on average 24 months.
  all the needs expressed by cancer patients and the related social-healthcare actions implemented will be recorded. To evaluate the feasibility of the social-healthcare pathway we will record the actions implemented successfully as well as the actions not implemented or ineffective.

SECONDARY OUTCOMES:
difficulties faced by cancer patients in the return to work process, collected by a guided interview (Feasibility indicator_2). | through study completion, on average 24 months.
  the difficulties arising from the guided interview will be analyzed qualitatively and categorized into emerging themes.
ratio of cancer patients who have returned to work/not returned to work (Feasibility indicator_3). | through study completion, on average 24 months.
  we will calculate the ratio among cancer patients who received only information support and among those who received information support and occupational therapy.
number of healthcare providers directly informed about UNAMANO (Feasibility indicator_4). | through study completion, on average 24 months.
  during the project, training events and meetings were organized with the aim to inform all the healthcare professionals of the AUSL-IRCCS of Reggio Emilia involved in the care and management of cancer patients about UNAMANO project.
number of healthcare professionals who refer patients to UNAMANO (Feasibility indicator_5). | through study completion, on average 24 months.
  during the project, training events and meetings were organized with the aim to inform all the healthcare professionals of the AUSL-IRCCS of Reggio Emilia involved in the care and management of cancer patients about UNAMANO project.
number of individuals that contact In-Forma Salute to seek information regarding UNAMANO without being referred by a healthcare professional (Feasibility indicator_6). | through study completion, on average 24 months.
  we have distributed flyers in the hospitals throughout the Province, launched the website of the project and published news in local and national newspapers and on social media in order to raise awareness and provide information to the local community regarding UNAMANO.
number of volunteers informed about UNAMANO and recruited by UNAMANO (Feasibility indicator_7). | through study completion, on average 24 months.
  we organize training events to recruit volunteers willing to support UNAMANO project.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Mazzini, Principal Investigator — Local Helath Authority of Reggio Emilia-IRCCS
Locations (1):
- Local Health Authority of Reggio Emilia-IRCCS, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paltrinieri S, Fugazzaro S, Bertozzi L, Bassi MC, Pellegrini M, Vicentini M, Mazzini E, Costi S. Return to work in European Cancer survivors: a systematic review. Support Care Cancer. 2018 Sep;26(9):2983-2994. doi: 10.1007/s00520-018-4270-6. Epub 2018 May 29. PMID 29845421
- [Background] Paltrinieri S, Vicentini M, Mazzini E, Ricchi E, Fugazzaro S, Mancuso P, Giorgi Rossi P, Costi S. Factors influencing return to work of cancer survivors: a population-based study in Italy. Support Care Cancer. 2020 Feb;28(2):701-712. doi: 10.1007/s00520-019-04868-0. Epub 2019 May 25. PMID 31129762